CLINICAL TRIAL: NCT04431323
Title: ESPRIMO: A Bio-psycho-social Co-created Intervention for Young Adults With Multiple Sclerosis: Study Protocol for a Feasibility Study
Brief Title: Intervention for Young Adults With Multiple Sclerosis
Acronym: ESPRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2676CESC
Record Dates: First submitted 2020-05-13; First posted 2020-06-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
Keywords: quality of life; young adults; biopsychosocial intervention
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: ESPRIMO is a feasibility study using a participatory design.
  It is composed of a pre-phase and three main consequential phases:
  * Pre-phase: Exploring the psychological impact of COVID-19 on young adults with MS using a cross-sectional web-based survey for patients with MS;
  * Phase 1 (Co-creation of the intervention): initial co-creation phase aiming to develop a biopsychosocial intervention (the so-called ESPRIMO intervention) targeted at young adults with MS, using cross-sectional web-based surveys for young adults with MS and healthcare providers as well as focus groups with patients;
  * Phase 2 (intervention): aiming to test preliminary effect, feasibility, and acceptability of the ESPRIMO intervention in a sample of young patients with MS; Phase 3 (Fine tuning of the intervention): evaluation of the results by the ESPRIMO Board (composed of four young adults with MS and three healthcare professionals) and subsequent fine-tuning of the ESPRIMO intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biopsychosocial intervention (Experimental): Young adults with MS will receive an intervention (group setting) composed of physical activities (duration: 10-12 weeks; either dancing or walking) and psychosocial interventions (6-8 encounters).
  [The intervention will start as soon as 8-10 patients will have been enrolled. A waiting list will be then created and patients contacted when the subsequent group starts. This waiting list does not serve as control group.
  One or more groups, respectively for the psychological intervention and the physical activities, may start at the same time but on different days, considering also the results of the co-creation phase.]
  Interventions: Behavioral: ESPRIMO

INTERVENTIONS:
Behavioral: ESPRIMO — Participants will receive the intervention during Phase 2.
  The intervention is based on the cognitive behavioral, the third-wave (mindfulness and acceptance and commitment therapy), and the positive psychology approach.
  The frequency of the intervention and the specific content and aims of the psychological and physical intervention will be based on the results of the surveys and the focus group discussion (Pre-phase and Phase 1). In order to maximize the benefit of the integrated intervention, all the three components of the interventions (i.e., psychological, motor exercise and social components) will be administered in the same time period.
  A preliminary theoretical framework of the intervention will be created prior to the survey phase according to the literature in the field. Specific aspects of this preliminary framework will be discussed during the co-creation phase and adapted after the analysis of the qualitative results.

SUMMARY:
This study aims to develop - in collaboration with patients with multiple sclerosis (MS)- a psychosocial and physical activity intervention (i.e., ESPRIMO intervention) for young adults with MS targeted at improving patients' health-related quality of life (HRQoL). Further, the study seeks to preliminarily test the effect, feasibility, and acceptability of the ESPRIMO intervention using a pilot sample of young adults with MS.

Given that the ESPRIMO study will be conducted immediately after the COVID-19 emergency, it does not seem reasonable to start the co-creation of the intervention without taking into account the potential impact of this pandemic on the quality of life and well-being of patients with MS and on their management of care. Thus, the investigators seek to better understand the needs of the target population under these particular circumstances.

DETAILED DESCRIPTION:
Being the most common neurological disease causing disability in young adults, multiple sclerosis (MS) does not only impair physical functions but is also often associated with fatigue, symptoms of depression and anxiety as well as reduced health related quality of life (HRQoL). Especially the first years after the diagnosis can be emotionally challenging and psychological adjustment problematic. Since MS is generally detected between the ages of 20 and 40, a period of great significance for professional and personal development, the adaptation to this chronic disease may become even more challenging.

It is now well established that psychological interventions aiming to support people with MS (e.g., Cognitive Behavioural Therapy, mindfulness-based interventions) do not only have a positive effect on psychological aspects, such as resilience, but also on physiological outcomes (e.g., fatigue, physical vitality) and on the perception of general health.

According to the literature, psychological well-being and HRQoL can be also promoted by regular physical activity and exercise (e.g., walking, ballroom dancing), which present the additional advantage of reducing some physical symptoms of MS. Practicing physical activity in groups enables participants also to socialize and create interpersonal relationships, which in turn may significantly affect patients' psychological well-being and illness perception.

Despite the positive impact of interventions focusing on either physical, psychological or social/interpersonal dimensions, there has been little discussion about the development of comprehensive interventions based on the bio-psycho-social model of disease. Even less attention has been paid to the development of early interventions tailored to young adults' needs and to the engagement of patients in the creation of such programs despite the fact that patient engagement has become a central priority for researchers and policy makers in medicine.

Therefore, the investigators aim to develop - in collaboration with patients with MS - a psychosocial and motor intervention (i.e., ESPRIMO intervention) for young adults with MS targeted at improving patients' HRQoL. Further, the study seeks to preliminarily test the effect, feasibility, and acceptability of the ESPRIMO intervention using a pilot sample of young adults with MS.

In the so-called co-creation phase, the primary aim is to create, together with patients, a bio-psycho-social intervention, following also the preferences and suggestions of healthcare professionals. In the intervention phase, the primary aim is to explore the feasibility of the intervention and its effect in improving their quality of life.

Secondary aims of the study are five-fold: 1) to collect patients' opinions and needs as well as healthcare professionals' perspectives on the preferred characteristics of a bio-psycho-social intervention; 2) to explore the effect of the bio-psycho-social intervention in improving bio-psycho-social aspects, such as quality of life, resilience, fatigue (see primary and secondary outcomes) 3) to investigate potential relationships between these psychological variables at baseline and post-intervention; 4) to assess the differences in effect, patient satisfaction and participation rates according to sociodemographic and clinical characteristics; 5) to examine the reasons for dropouts and possible barriers to participation.

Additionally, considering that the ESPRIMO Study will start shortly after the end of the COVID-19 emergency, the potential impact of this emergency on patients' well-being and quality of life must be taken into account when creating the intervention together with the patients.

Therefore, the investigators aim to explore in a pre-phase the potential impact of the COVID-19 emergency on the psychological status and management of disease and the potential positive resources used to deal with this highly challenging situation.

ELIGIBILITY:
As different samples of patients and healthcare professionals will be enrolled in the different phases of the studies, inclusion and exclusion criteria vary:

1. Explorative pre-phase "Exploring the psychological impact of the COVID-19 emergency"

   Inclusion Criteria:
   * age range: 18-45 years;
   * MS Diagnosis;
   * Italian speakers;
   * electronic informed consent signed.

   Exclusion Criteria:
   * N/A
2. Co-creation phase - Survey with young adults with MS

   Inclusion Criteria:
   * age range: 18-45 years;
   * MS diagnosis;
   * Italian speakers;
   * electronic informed consent signed.

   Exclusion Criteria:

   -N/A
3. Co-creation phase - Survey with Healthcare Providers

   Inclusion Criteria:
   * being a healthcare professional working with MS patients;
   * Italian speakers;
   * electronic informed consent signed.

   Exclusion Criteria:

   -N/A
4. Co-creation phase - Focus groups

   Inclusion Criteria:
   * age range: 18-45 years;
   * MS diagnosis;
   * Italian speakers;
   * signed informed consent.

   Exclusion Criteria:

   -N/A
5. Intervention phase

Inclusion Criteria:

* age range: 18-45 years;
* Ms diagnosis according to the revised McDonald Criteria [Thompson et al., 2018];
* Italian speakers;
* Signed informed consent.

Exclusion Criteria:

* clinically relevant cognitive deficits as evaluated by the treating neurologist which may represent obstacles in filling the questionnaires and participating in the intervention;
* severe psychiatric disorders, such as psychosis, bipolar disorder, active substance abuse problems, dissociative disorders, or a current diagnosis of major depression as evaluated by the neurologist or the clinical psychologist;
* clinically relevant physical impairments rendering impossible the physical activities included in the intervention, defined as an Expanded Disability Status Scale (EDSS) score higher than 3.5 [Bowen et al., 2001].

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Health-related Quality of Life up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Health-related Quality of Life at 1 day post-intervention will be Health-related quality of life will be measured by the Italian version of the "Coop/Wonca charts" [van Weel et al., 1993] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The Coop/Wonca questionnaire is a self-reported single-item scale to explore HRQoL, including physical (fitness and daily activities), mental (emotions), social domains (social contacts) and above that general health and change in health status [Weel et al., 1995]. Each chart consists of a single question referring to the preceding two weeks and are scored on a 5-level ordinal scale ranging from 1 (no impact) to 5 (high impact), illustrated by a simple picture.
Acceptance and Satisfaction with the Intervention assessed by an ad hoc questionnaire | T1: up to 1 week post-intervention
  An ad hoc questionnaire (one of the two specific outcome measures evaluating the feasibility of the intervention) using closed (rated by Likert scales ranging from 1 (not at all) to 10 (very much, with higher scores reflecting higher levels of acceptance and satisfaction) and open questions will be administered to evaluate the acceptance and satisfaction of participants.
  Information on participants' experience will inform the intervention and its administration and will reduce barriers to participation for future patients.

SECONDARY OUTCOMES:
Change from Baseline Resilience Features up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Resilience will be measured using the Italian version of the "Connor-Davidson Resilience Scale" [CD-RISC; Connor & Davidson, 2003] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The CD-RISC is designed to assess resilience features in adolescents and adults and composed of 25 items and evaluated on a 5-point Likert scale (ranging from 0 "not true at all" to 4 "true nearly all of the time"), with higher scores reflecting higher levels of resilience.
Change from Baseline Well-being up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Well-being will be measured using the Italian version of the "Short Form 12 general health questionnaire" [SF12, Apolone et al., 2001] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The SF12 is a validated 12-item questionnaire with Physical and Mental Component Summary (PCS and MCS, respectively) scores.
  The SF12 uses different types of scales (e.g., Yes/No questions, scales ranging from 1(always) to 6 (never)).
Change from Baseline Mindfulness Traits up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Mindfulness traits will be assessed using the Italian version of the "Five Facet Mindfulness Questionnaire" [FFMQ; Baer et al., 2006; Giovannini et al., 2014] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The FFMQ-SF is a 24-item self-report questionnaire measuring one general mindfulness factor and five secondary facets (i.e., Observe, Describe, Act with Awareness, Nonjudge, and Nonreact) on a 5-point Likert scale, ranging from 1 ("never or very rarely true") to 5 ("very often or always true"), with higher total scores reflecting a greater degree of mindfulness.
Change from Baseline Self-efficacy in MS up to 1 week post-intervention assessed by the "Self-Efficacy in Multiple Sclerosis Scale" (SEMS) | T0: baseline, T1: up to 1 week post-intervention
  Self-efficacy will be measured using the "Self-Efficacy in Multiple Sclerosis Scale" [SEMS; Bonino et al., 2016] at baseline and 1 day post-intervention assessing the changes between the two time points.
  It is a 15-item self-completion instrument using a 5-point Likert scale (from 0 = not at all confident to 4 = very confident). Items are conceptually allocated to two areas: "Goal setting" (9 items) and "Symptom management" (6 items).
Change from Baseline Perceived Social Support up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Perceived social support will be measured using the "Multidimensional Scale of Perceived Social Support" [MSPSS; Prezza & Principato, 2002; Zimet et al., 1988] at baseline and 1 day post-intervention assessing the changes between the two time points.
  It is a 12-item self-report measure, assessing on a 7-point Likert scale (from 1 "strongly disagree" to 7 "strongly agree") the level of perceived social support of various sources: family, friends, and significant others.
Change from Baseline Levels of Anxiety and Depression up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Levels of anxiety and depression will be measured using the "Hospital Anxiety and Depression Scale" [HADS; Zigmond & Snaith, 1983; Costantini et al., 1999] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The HADS is a brief self-report questionnaire composed of 14 items describing on a 4-point scale from 0 to 3 the levels of anxiety a person is experiencing.
  HADS anxiety (HADS-A, 7 items) and depression (HADS-D, 7 items) subscale scores will be calculated, possibly ranging from 0 (no symptoms) to 21 (most severe symptoms). A HADS-A and HADS-D score of ≥8 indicates a high risk of anxiety and depressive disorder.
Change from Baseline Illness Representations up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Illness perception will be measured using the "Brief Illness Perception Questionnaire" [Brief IPQ-R; Broadbent et al., 2006; Pain et al., 2006] at baseline and 1 day post-intervention assessing the changes between the two time points.
  It is a 9-item self-completion instrument using a 5-point Likert scale (from "strongly disagree" to "strongly agree") providing a quantitative measurement of the components of illness representations [Leventhal et al., 1984; Leventhal et al., 1997].
Change from Baseline Committed Action up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  The construct of committed action is measured applying the Italian version of the "The Committed Action Questionnaire-8" (CAQ-8) [McCracken et al., 2015] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The CAQ-8, a short version of The Committed Action Questionnaire [McCracken, 2013], is an 8-item questionnaire using a 7-point Likert scale (from 0 = never true to 6 = always true).
Change from Baseline Levels of (Motor and Cognitive) Fatigue up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Fatigue will be measured applying the "Fatigue Scale for Motor and Cognitive Functions" [FSMC; Penner et al., 2009; Elbers et al., 2012] at baseline and 1 day post-intervention assessing the changes between the two time points.
  It is a self-report fatigue questionnaires validated in patients with multiple sclerosis (MS) and useful to evaluate both motor and cognitive fatigue.
  It is composed by 20 items evaluated on a Likert scale, ranging from 1 (it never happens) to 5 (it always happens), with higher scores reflecting higher levels of motor and cognitive fatigue.
Change from Baseline Perceived Autonomy Support up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Perceived autonomy support (as part of a set of variables reflecting attitudes towards physical activity and motivation to be physically active) will be measured with the "Perceived Autonomy Support Scale for Exercise Setting" (PASSES; Hagger et al., 2007) at baseline and 1 day post-intervention assessing the changes between the two time points.
  The 12 items are rated on a 7-point Likert scale ranging from 1(totally disagree) to 7 (totally agree), with higher scores reflecting greater perceptions of autonomy support.
Change from Baseline Autonomous Motivation up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Autonomous motivation (as part of a set of variables reflecting attitudes towards physical activity and motivation to be physically active) will be measured with the "Behavioral Regulation in Exercise Questionnaire" [BREQ-3; Markland et al., 2014] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The 24 items are rated on a 5-point Likert scale ranging from 1 (totally disagree) to 5 (totally agree).
Change from Baseline Attitudes up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Attitudes (as part of a set of variables reflecting attitudes towards physical activity and motivation to be physically active) will be measured by a scale developed by Galli et al. [2018], following the recommendations of Ajzen [1991] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The scale comprises 6 items with responses provided on seven-points scales (with contrasting adjectives (e.g.,"bad - good", "harmful-beneficial").
Change from Baseline Subjective Norms up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Subjective norms (as part of a set of variables reflecting attitudes towards physical activity and motivation to be physically active) will be measured by a scale developed by Galli et al. [2018], following the recommendations of Ajzen [1991] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The 3 items of the scale are rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree), with a greater single score (aggregated item scores) indicating greater normative social pressure toward the behavior.
Change from Baseline Perceived Behavioral Control up to 1 week post-intervention | T0: baseline, T1: up to 1 week post-intervention
  Perceived Behavioral Control (as part of a set of variables reflecting attitudes towards physical activity and motivation to be physically active) will be measured by a scale developed by Galli et al. [2018], following the recommendations of Ajzen [1991] at baseline and 1 day post-intervention assessing the changes between the two time points.
  The 3 items of the scale are rated on a 7-point Likert scale, with a greater single score (aggregated item scores) indicating greater perceived confidence toward the behavior.
Change from baseline number of steps/day to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the number of steps/day.
Change from baseline km traveled/day to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the number of km traveled/day.
Change from baseline number of active hours/day to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the number of active hours/day.
Change from baseline number of inactive hours/day to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the number of inactive hours/day.
Change from Baseline number of hours of sleep/day to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the number of hours of sleep/day.
Change from baseline heart rate to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the heart rate (HR).
Change from baseline heart rate variability to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the heart rate variability (HRV).
Change from estimated kilocalories consumed/day at baseline to 5 days post-intervention | T0: baseline, T1: 5 days post-intervention
  A smartwatch will be used by each patient for 5 days at baseline (T0) and 5 days after the intervention (T1) in order to compare the estimated kilocalories consumed/day.
Number of Drop Outs | T1: up to 1 week post-intervention
  The number of drop outs is the second specific outcome measure evaluating the feasibility of the intervention.
Exact Time of Dropping Out | T1: up to 1 week post-intervention
  The exact time point of dropping out will also be assessed.
Underlying Reasons for Dropping Out assessed by an ad hoc questionnaire with open questions | T1: up to 1 week post-intervention
  Patients who drop out during the interventions will be contacted to assess the underlying reasons using an ad hoc questionnaire with open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Rimondini, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Alberto Gajofatto Study Principal Investigator, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Policlinico G.B. Rossi, Verona, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for the primary and secondary outcome measures will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data can be made available upon reasonable request when data are published (6 months after publication).
Access Criteria: Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Bowen J, Gibbons L, Gianas A, Kraft GH. Self-administered Expanded Disability Status Scale with functional system scores correlates well with a physician-administered test. Mult Scler. 2001 Jun;7(3):201-6. doi: 10.1177/135245850100700311. PMID 11475445
- [Background] Van Weel C. Functional status in primary care: COOP/WONCA charts. Disabil Rehabil. 1993 Apr-Jun;15(2):96-101. doi: 10.3109/09638289309165878. PMID 8513163
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Apolone G, Mosconi P, Quattrociocchi L, et al. Questionario sullo stato di salute SF-12. Versione italiana. Milano: Guerini e Associati, 2001.
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Giovannini C, Giromini L, Bonalume L, et al. The Italian Five Facet Mindfulness Questionnaire: A Contribution to its Validity and Reliability. J Psychopathol Behav Assess 2014; 36.doi: 10.1007/s10862-013-9403-0.
- [Background] Bonino S, Graziano F, Borghi M, et al. The Self-Efficacy in Multiple Sclerosis (SEMS) Scale: Development and Validation With Rasch Analysis. European Journal of Psychological Assessment. 2015; doi: 10.1027/1015-5759/a000350.
- [Background] Costantini M, Musso M, Viterbori P, Bonci F, Del Mastro L, Garrone O, Venturini M, Morasso G. Detecting psychological distress in cancer patients: validity of the Italian version of the Hospital Anxiety and Depression Scale. Support Care Cancer. 1999 May;7(3):121-7. doi: 10.1007/s005200050241. PMID 10335929
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Pain D, Miglioretti M, Angelino, E. Development of Italian version of brief-IPQ (Illness perception questionnaire, short version), a method for assessing the illness representations. Psicologia della Salute. 2006. 81-89.
- [Background] Leventhal H, Nerenz DR, Steele DS. Illness representations and coping with health threats. In: Baum, A. Taylor, S.E. and Singer, J.E. (Eds.), Handbook of psychology and health. Vol. IV. pp. 219-252. Hillsdale, NJ: Erlbaum, 1984.
- [Background] Leventhal H, Benyamini Y, Brownlee S, et al. Illness representations: Theoretical foundations. In K. J. Petrie & J. A. Weinman (Ed.), Perceptions of health and illness: Current research and applications (p. 19-45). Reading, UK: Harwood Academic Publishers, 1997.
- [Background] McCracken LM. Committed action: an application of the psychological flexibility model to activity patterns in chronic pain. J Pain. 2013 Aug;14(8):828-35. doi: 10.1016/j.jpain.2013.02.009. Epub 2013 May 4. PMID 23651881
- [Background] McCracken LM, Chilcot J, Norton S. Further development in the assessment of psychological flexibility: a shortened Committed Action Questionnaire (CAQ-8). Eur J Pain. 2015 May;19(5):677-85. doi: 10.1002/ejp.589. Epub 2014 Sep 2. PMID 25181605
- [Background] Penner IK, Raselli C, Stocklin M, Opwis K, Kappos L, Calabrese P. The Fatigue Scale for Motor and Cognitive Functions (FSMC): validation of a new instrument to assess multiple sclerosis-related fatigue. Mult Scler. 2009 Dec;15(12):1509-17. doi: 10.1177/1352458509348519. Epub 2009 Dec 7. PMID 19995840
- [Background] Elbers RG, Rietberg MB, van Wegen EE, Verhoef J, Kramer SF, Terwee CB, Kwakkel G. Self-report fatigue questionnaires in multiple sclerosis, Parkinson's disease and stroke: a systematic review of measurement properties. Qual Life Res. 2012 Aug;21(6):925-44. doi: 10.1007/s11136-011-0009-2. Epub 2011 Oct 20. PMID 22012025
- [Background] Prezza M, Principato MC. La rete e il sostegno sociale. In: Prezza M, Santinello M, eds. Conoscere la comunit . Bologna. Italy: Il Mulino, 2002: 193-233.
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991;50:179- 211.
- [Background] Galli F, Chirico A, Mallia L, Girelli L, De Laurentiis M, Lucidi F, Giordano A, Botti G. Active lifestyles in older adults: an integrated predictive model of physical activity and exercise. Oncotarget. 2018 May 22;9(39):25402-25413. doi: 10.18632/oncotarget.25352. eCollection 2018 May 22. PMID 29875997
- [Derived] Poli S, Donisi V, Mazzi MA, Gobbin F, Giusto G, Orlandi R, Schena F, Del Piccolo L, das Nair R, Gajofatto A, Rimondini M. Fostering quality of life in young adults living with multiple sclerosis: a pilot study of a co-created integrated intervention. Front Psychol. 2024 Mar 26;15:1342166. doi: 10.3389/fpsyg.2024.1342166. eCollection 2024. PMID 38596329